CLINICAL TRIAL: NCT06888154
Title: The Effect of Hot Compress Applied on the Intestines on Postoperative Nausea-vomiting and Bowel Function in Abdominal Surgery
Brief Title: Hot Compress Application in Open Abdominal Surgery
Acronym: HotCompress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Dilek Talhaoglu, Assistant Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: hot compress
Record Dates: First submitted 2025-03-09; First posted 2025-03-21 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Abdominal Surgery by Laparotomy
Keywords: abdominal surgery; hot compress; operating room; nursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Hot compress Application) (Experimental): Patients in this group will be toweled with heated saline during abdominal surgery. After the abdomen is opened, the intestines will be covered with a sterile towel soaked in saline heated to 36°C to prevent drying and reduce the risk of infection.
  Interventions: Other: compress application with heated saline
- Control Group (Routine Care) (No Intervention): Patients in this group will receive standard surgical care.

INTERVENTIONS:
Other: compress application with heated saline — Covering intestines with sterile gauze soaked in 36°C heated saline during surgery to prevent drying and reduce infection risk
  Arms: Intervention Group (Hot compress Application)

SUMMARY:
This study aims to evaluate the effect of hot compress application to the intestines during abdominal surgery on postoperative nausea-vomiting and bowel function.

Volunteers will be randomly assigned to the intervention and control groups. Initially, 30 patients will be included in each group, and the study will be completed based on the effect size determined by power analysis.

Hypotheses:

H0: Covering the intestines with saline heated at 36°C during surgery has no effect on postoperative nausea and vomiting.

H1: Covering the intestines with saline heated at 36°C during surgery affects postoperative nausea and vomiting.

H01: Covering the intestines with saline heated at 36°C during surgery has no effect on postoperative bowel function.

H11: Covering the intestines with saline heated at 36°C during surgery affects postoperative bowel function.

Inclusion Criteria:

Undergoing abdominal surgery in the general surgery ward, Aged 18 years or older, Having a BMI between 18.50-24.99 kg/m², Able to communicate verbally, Willing to participate in the study, Conscious and oriented patients.

Exclusion Criteria:

History of previous gastrointestinal surgery, Postoperative complications, History of small bowel resection, ileostomy, or colostomy, History of emergency surgery, neoadjuvant therapy, appendectomy, or inflammatory bowel disease, Chronic opioid use, Chronic constipation (≤ 2 bowel movements per week), History of abdominal radiotherapy, Admission to the intensive care unit or postoperative bleeding.

Application:

Intervention Group: Routine preoperative procedures will be performed. During surgery, the intestines will be covered with sterile gauze soaked in saline heated at 36°C to prevent drying and reduce the risk of infection. Routine postoperative procedures will also be applied.

Control Group: Routine preoperative, intraoperative, and postoperative procedures will be applied. During surgery, the intestines will be covered with sterile gauze soaked in unheated saline, following standard practice.

Outcome Measures:

Primary Outcome: Gastrointestinal function assessment index, including time to first flatulence, first defecation, first normal bowel sounds, and first consumption of liquid/semi-solid food.

Secondary Outcome: Gastrointestinal symptoms such as nausea, abdominal bloating, pain, and vomiting.

DETAILED DESCRIPTION:
DATA COLLECTION Patient Introduction Form (ANNEX-1) and Patient Follow-up Form (ANNEX-2), Healing Quality-15 Scale (ANNEX-3) and Gastrointestinal Symptom Rating Scale (ANNEX-4), which were created by the researchers by reviewing the literature will be used for data collection.

Patient Introduction Form:

The Patient Information Form, which was created by the researchers by reviewing the literature includes questions about age, gender, medical diagnosis, educational status, BMI, chronic disease, medication used continuously, previous surgery, and frequency of defecation.

Patient Follow-up Form:

The Patient Introduction Form, which was created by the researchers by reviewing the literature , consists of 3 sections including preoperative, intraoperative and postoperative. In the preoperative section, preoperative lab. findings, preoperative fasting time (hours), type and amount of IV fluid given preoperatively; In the intraoperative section, surgical method, amount of fluid given in surgery, duration of surgery (min), fluid given in surgery, blood transfusion administration in surgery; In the postoperative section, laboratory findings, blood transfusion, presence of drain, pain, serum administered postoper

Quality Of Recovery-15 Scale/Quality Of Recovery-15 (QoR-15):

The QoR-15 scale is a validated tool used to assess postoperative recovery quality. It consists of 15 items, each scored on a 0-10 scale, with a total score range of 0 to 150 (higher scores indicate better recovery).

Gastrointestinal Symptom Rating Scale The GDSS (Gastrointestinal Symptom Rating Scale) is a 15-item, 7-point Likert-type scale with options ranging from "no discomfort" to "very severe discomfort".

The Gastrointestinal Symptom Rating Scale (GSRS) is a validated tool used to assess the severity of gastrointestinal (GI) symptoms. It consists of 15 items, each scored on a 7-point Likert scale (1 = no discomfort, 7 = severe discomfort).

Scoring Interpretation:

Total Score Range: 15 to 105 (higher scores indicate worse GI symptoms). Mean score calculation: Total score is divided by the number of items (15) to determine the severity of symptoms.

Interpretation of Scores:

15 - 30 → Mild symptoms 31 - 60 → Moderate symptoms 61 - 105 → Severe symptoms

ELIGIBILITY:
Inclusion Criteria:

* Abdominal surgery in the general surgery ward
* 18 years of age or older
* Patients with BMI in the normal range (18.50-24.99 kg/m2)
* Able to communicate verbally
* Those who volunteered to participate in the study
* Patients with no mental confusion, conscious and oriented will be included.

Exclusion Criteria:

* Previous gastrointestinal system surgery
* Complications in the postoperative period
* History of small bowel resection and ileostomy or colostomy
* Surgical history of inflammatory bowel diseases, emergency surgery, neoadjuvant therapy, appendectomy,
* Chronic opioid use,
* Experiencing chronic constipation (≤ 2 bowel movements per week),
* Abdominal radiotherapy
* Patients admitted to intensive care unit and patients with bleeding will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
will be an index of gastrointestinal functional assessment, including time to first passing gas, first defecation, first normal bowel sounds and first consumption of liquid/semi-general diet foods | postoperative 1-3 day
  Quality of Recovery-15 (QoR-15) Scale Scores:
  The QoR-15 scale is a validated tool used to assess postoperative recovery quality. It consists of 15 items, each scored on a 0-10 scale, with a total score range of 0 to 150 (higher scores indicate better recovery).
  Scoring Interpretation:
  0 - 70 → Poor recovery 71 - 100 → Moderate recovery 101 - 150 → Good recovery
  Gastrointestinal Symptom Rating Scale (GSRS) - Scale Scores The Gastrointestinal Symptom Rating Scale (GSRS) is a validated tool used to assess the severity of gastrointestinal (GI) symptoms. It consists of 15 items, each scored on a 7-point Likert scale (1 = no discomfort, 7 = severe discomfort).
  Scoring Interpretation:
  Total Score Range: 15 to 105 (higher scores indicate worse GI symptoms). Mean score calculation: Total score is divided by the number of items (15) to determine the severity of symptoms.
  Interpretation of Scores:
  15 - 30 → Mild symptoms 31 - 60 → Moderate symptoms 61 - 105 → Severe symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Merkez, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No